CLINICAL TRIAL: NCT00961363
Title: The Effect of Sitagliptin on Postprandial Glycemia and Endothelial Function in Chinese Subjects With Impaired Glucose Tolerance
Brief Title: Effect of Sitagliptin in Impaired Glucose Tolerance
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Professor Lee-Ming Chuang, National Taiwan Univerisity Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 200904052M
Record Dates: First submitted 2009-08-11; First posted 2009-08-18 (Estimated); Last update posted 2010-03-22 (Estimated); Status verified 2010-03

CONDITIONS: Impaired Glucose Tolerance
MeSH Terms: conditions — Glucose Intolerance | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin (Experimental): Sitagliptin
  Interventions: Drug: Sitagliptin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin — sitagliptin 100 mg per day
  Arms: Sitagliptin
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the safety and efficacy of sitagliptin 100 mg every day (q.d.) in improving hyperglycemia and endothelial dysfunction in subjects with impaired glucose tolerance.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese subjects aged 40-65 years with fasting plasma glucose < 100 mg/dL and OGTT 2-hour glucose 140-199 mg/dL.
2. Subjects are judged to be in otherwise general good health based on medical history, physical examination, and routine laboratory tests.
3. Subject has an understanding of the study procedures, alternative treatments available and risk involved with the study, and voluntarily agrees to participate by giving written informed consent.
4. Non-sterilized premenopausal female agrees to receive pregnancy test to confirm the non-pregnancy status and use adequate contraceptive methods to prevent pregnancy during the study period. Patient status should be confirmed by pregnancy test before enrollment.

Exclusion Criteria:

1. Evidence of diabetes (FPG> 125 mg/dL, or OGTT 2-hour glucose>=200 mg/dL, or current use of an anti-diabetic agents, except for history of gestational diabetes).
2. History of intolerance or hypersensitivity or contraindication as mentioned in the approved package insert (appendix).
3. Patient has any of the following disorders within the past 6 months: acute coronary syndrome (e.g., MI or unstable angina), coronary artery intervention (e.g., CABG or PTCA), stroke or transient ischemic neurological disorder.
4. Patient has new or worsening signs or symptoms of coronary heart disease within the past 3 months.
5. Patient has a BMI > 40 kg/m2.
6. Patient is on or likely to require more than 14 consecutive days or repeated courses of pharmacologic doses of corticosteroids. Note: inhaled, nasal, and topical corticosteroids are permitted.
7. Patient is on or likely to require treatment with immunosuppressive agents (e.g., cyclosporine, methotrexate).
8. Advanced renal insufficiency (estimated creatinine clearance < 50 ml/min).
9. Severe hepatic insufficiency (Child-Pugh score > 9, see Appendix).

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
the change in fasting and post-load plasma glucose levels during OGTT | 24 weeks

SECONDARY OUTCOMES:
the changes in endothelial function, measured by circulating adhesion molecules | 24 weeks
the changes in beta cell functions derived from the glucose/insulin levels during OGTT | 24 weeks
the safety and the tolerability of sitagliptin, including clinical and laboratory adverse experiences, laboratory values, weight, and vital signs. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lee-Ming Chuang, MD, PhD, Principal Investigator — Department of Internal Medicine, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan